CLINICAL TRIAL: NCT05694650
Title: Perceptions of Hospital Care at Home for Patients With Cancer: A Qualitative Study of Cancer Providers, Patients and Caregivers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0654; NCI-2022-09841 (Other: NCI CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus: Participants will be asked about your previous experiences providing cancer care at MD Anderson and your thoughts on providing hospital care at home
  Interventions: Behavioral: Focus Group; Behavioral: Interview
- Interview: Participants will be asked about your previous experiences providing cancer care at MD Anderson and your thoughts on providing hospital care at home
  Interventions: Behavioral: Focus Group; Behavioral: Interview

INTERVENTIONS:
Behavioral: Focus Group — Participants can meet with an interviewer alone. The focus group should take about 1 hour and will be held in person at MD Anderson, by telephone, or online using a video conferencing app called Zoom
Behavioral: Interview — Participants can meet with an interviewer alone. The interview should take about 1 hour and will be held in person at MD Anderson, by telephone, or online using a video conferencing app called Zoom

SUMMARY:
The objective of this qualitative research study is to assess the knowledge, attitudes and beliefs of cancer care providers, patients with cancer and caregivers regarding hospital care at home. We aim to conduct qualitative interviews to inform implementation of future on oncology hospital care at home programs

DETAILED DESCRIPTION:
Interviews and focus groups will be conducted in English only using an interview guide (attached). The interview guide was based on the Consolidated Framework for Implementation Research (CFIR)8 to provide a broad understanding of the potential barriers and enablers of implementing a hospital care at home program. In summary, interviews will begin with an overview of the qualitative research study followed by verification of a completed demographic questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Cancer Care Providers

   * Cancer care providers of any specialty, including but not limited to oncologists, surgeons, hospitalists, emergency medicine physicians, nurses (including nurse practitioners), physician assistants, and any other member of the cancer care team (eg social workers or physical therapists)
   * Employed by the University of Texas MD Anderson Cancer Center
2. Patients

   * Adults ages 18 and over
   * Currently undergoing or completed cancer treatment within the last 5 years at MD Anderson
   * Able to speak and read in English
3. Caregivers

   * Adults ages 18 and over
   * Self-identifies as a caregiver of an individual over 18 who is currently undergoing cancer treatment or completed cancer treatment within the last 5 years at MD Anderson
   * Able to speak and read in English

Exclusion:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaires | through study completion an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tacara Soones, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org